CLINICAL TRIAL: NCT03533946
Title: A Phase II Study of Rucaparib Monotherapy in Nonmetastatic, Hormone-Sensitive Prostate Cancer Demonstrating "BRCAness" Genotype (ROAR)
Brief Title: Rucaparib in Nonmetastatic prOstAte With BRCAness
Acronym: ROAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: New standard of care for study participant population
Sponsor: University of Utah (Other)
Collaborators: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI111833
Record Dates: First submitted 2018-04-26; First posted 2018-05-23 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — rucaparib

STUDY DESIGN:
Intervention Model Description: This is a single arm, open label, phase II trial to assess efficacy of rucaparib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rucaparib, all participants (Experimental): Single Arm study, all participants will get rucaparib
  Interventions: Drug: Rucaparib

INTERVENTIONS:
Drug: Rucaparib — Treatment with rucaparib will begin on Cycle 1 Day 1 and continue at 600 mg twice daily. Therapy continues until Prostate Specific Antigen (PSA) progression or intolerable toxicities.
  Other Names: Rubraca

SUMMARY:
This is a single arm, open label, phase II trial to assess efficacy of rucaparib.

ELIGIBILITY:
Inclusion Criteria:

* Hormone-sensitive, histologically proven adenocarcinoma of the prostate with BRCAness (defined as an alteration in one or more of the following genes: BARD1, BRCA1, BRCA2, BRIP1, CHEK1, CHEK2, FANCA, NBN, PALB2, RAD51C, RAD51D, RAD51, RAD51B) from soft-tissue based genomic testing or liquid biopsy based genomic or genetic testing. Pathogenic or likely pathogenic alterations are accepted.
* Eastern Cooperative Oncology Group (ECOG)/Zubrod score of 0-2.
* At a minimum, subjects must have received definitive local therapy with curative intent (i.e., prostatectomy, and/or radiation therapy) with or without systemic therapy.
* Testosterone level is > 50 ng/dL.
* Be at least 18 years old at the time the informed consent form is signed.
* Demonstrate adequate organ function as defined in the table in the protocol, all screening labs should be performed within 28 days of treatment initiation.
* Highly effective barrier methods must be used with all sexual activity and contraception methods must be practiced for all subjects throughout the study and for at least 6 months after last rucaparib treatment administration if the risk of conception exists (section 7.2).
* Recovery to baseline or Grade ≤ 1 CTCAE v5.0 from toxicities related to any prior treatments within the context of their definitive local therapy for their prostate cancer, unless Adverse Event(s) (AE)(s) are clinically nonsignificant and/or stable on supportive therapy.
* Subject is able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Subject must have confirmed PSA progression based on at least two time points taken at least one week apart to confirm rising trend.

Exclusion Criteria:

* Subjects with metastases defined by conventional scans (CT, MRI, Nuclear Medicine (NM) Bone Scan). Disease identified on molecular imaging (e.g. fluciclovine-PET) is not exclusionary.
* Arterial or venous thrombi (including cerebrovascular accident), myocardial infarction, admission for unstable angina, cardiac angioplasty, or stenting within the last 90 days prior to screening.
* Pre-existing duodenal stent, recent (within < 3 months) or existing bowel obstruction, and/or any gastrointestinal disorder or defect that would, in the opinion of the Investigator, interfere with absorption of rucaparib.
* Inability to swallow tablets.
* Evidence or history of clinically significant bleeding disorder per the determination of the treating investigator.
* Prior systemic therapy within the past 30 days prior to Day 1 (or 5 half-lives of the drug, whichever is shorter).
* Diagnosis of another malignancy within 2 years before first dose of study treatment only if the cancer will either interfere with participant safety or interfere with the primary endpoint, per the judgement of the Principal Investigator. Participants, who have been diagnosed with, superficial skin cancers, or localized, low grade tumors deemed cured or with a prolonged natural history (e.g estimated overall survival > 5 years) may be included.
* Prior treatment with any poly adenosine diphosphate-ribose polymerase (PARP) inhibitor, mitoxantrone, cyclophosphamide, or any platinum based chemotherapy.
* Clinically significant (i.e., active) cardiovascular disease at the time of enrollment: congestive heart failure (> New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Other severe acute or chronic medical conditions including cardiovascular, endocrine, neurologic, pulmonary or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before first dose and from minor surgery (eg, simple excision, tooth extraction) at least 28 days before first dose. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahu KK, Li H, Mathew Thomas V, Benson M, Boucher K, Gupta S, Kohli M, Swami U, Agarwal N, Maughan BL. A Phase II Study of Rucaparib Monotherapy in Nonmetastatic, Hormone-Sensitive Prostate Cancer Demonstrating "BRCAness" Genotype (ROAR). Oncologist. 2024 May 3;29(5):450-e725. doi: 10.1093/oncolo/oyae030. PMID 38452035

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rucaparib, All Participants
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rucaparib, All Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Age, Continuous [Median (Standard Deviation); unit: years] | 69 (5.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen Progression Free Survival
Description: The levels of PSA were monitored monthly for comparison to baseline levels until the time of PSA progression, or 2 years after study treatment discontinuation, or study termination, as defined by Prostate Cancer Working Group 3 (PCWG3) criteria. PCWG3 criteria for PSA progression is a rise over baseline of >= 25% and an absolute rise of >= 2 ng/mL. Reported as median number of months from baseline to PSA progression.
Time Frame: From baseline to up to 2 years after study treatment discontinuation; actual max approximately 42 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rucaparib, All Participants
Number analyzed (Participants) | 7
Months | 35.37 [0 to 85.11]

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) Related to Rucaparib
Description: To assess the safety of rucaparib in participants with biochemically recurrent hormone-sensitive prostate cancer.
  Severity of adverse events was assessed using CTCAE v5.0 criteria, a 1-5 scale with higher numbers indicating greater severity, where Grade 1 indicates "mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated" and Grade 5 indicates "death related to AE." Each adverse event was also evaluated by the treating investigator to assess its attribution to rucaparib, with options being unrelated, unlikely related, possibly related, probably related, or definitely related to rucaparib. Possibly, probably, and definitely related were grouped together as "Related." Reported here are the number of participants with any related AE of the specified grade. Note that there were no Grade 4 or Grade 5 related AEs.
Time Frame: From first dose of study treatment until 30 days after last dose of study treatment; max 42 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib, All Participants
Number analyzed (Participants) | 7
Participants
  Grade 1 | 7
  Grade 2 | 4
  Grade 3 | 2

3. Secondary Outcome: Count of Participants With an Undetectable PSA at 6 and 12 Months
Description: To assess the percentage of participants with an undetectable PSA after initiation of study therapy at 6 and 12 months.
  Endpoint: the levels of PSA will be monitored monthly for comparison to baseline levels to determine when PSA becomes undetectable. Participants who were not followed for at least 6 months after initiation of study therapy were not able to be evaluated for this time point.
Time Frame: At 6 and 12 months after initiation of study therapy
Population: Three participants did not complete follow-up to 6 months, so only four could be evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib, All Participants
Number analyzed (Participants) | 4
Participants
  At 6 months | 1
  At 12 months | 1

4. Secondary Outcome: Overall Survival (OS) at 2 Years
Description: To evaluate OS in nonmetastatic hormone-sensitive prostrate cancer participants treated with rucaparib. Calculated as the number of participants alive 2 years after study treatment discontinuation or study termination.
Time Frame: From start of study treatment until up to 2 years after study treatment discontinuation; actual max approximately 42 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib, All Participants
Number analyzed (Participants) | 7
Participants | 7

5. Secondary Outcome: Count of Participants With 50% or Greater Reduction in PSA Levels
Description: To assess the number of participants with a 50% reduction in PSA levels (PSA50) compared to the baseline value at the time of study enrollment. The levels of PSA will be monitored monthly for comparison to baseline levels.
Time Frame: From baseline until up to 2 years after study treatment discontinuation; actual max approximately 42 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib, All Participants
Number analyzed (Participants) | 7
Participants | 2

ADVERSE EVENTS:
Time Frame: From start of study treatment until 30 days after discontinuation of study treatment; max approximately 42 months
Description: Adverse events were assessed at each study visit (approximately monthly). The occurrence of adverse events was sought by non-directive questioning of the participant at each visit or phone contact during the study. Adverse events also may have been detected when they were volunteered by the participant during or between visits or through physical examination, laboratory test, or other assessments.
Arm/Group | Rucaparib, All Participants
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rucaparib, All Participants (N=7)
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 2
Bloating (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 5 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 — Barrett's Esophagus (1); Blood in Stool (1)
Headache (Nervous system disorders) | 2
Hematoma (Vascular disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 — Ingrown Hair (1)
Insomnia (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Localized edema (General disorders) | 1
Memory impairment (Nervous system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — Compressed Lumbar Disc (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Cyst (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Decreased Pain Recognition (1)
Oral dysesthesia (Gastrointestinal disorders) | 1
Otitis externa (Infections and infestations) | 1
Pain (General disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Presyncope (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (2) — Panic Attacks (1); Vivid Dreams (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Blistering (1)
Skin infection (Infections and infestations) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 4 (11) — Cataract Lens Replacement (1); Colonoscopy (2); Cyst Removal (1 participant, 2 events); Endoscopy (1); Eye Surgery (1); Inspire Implant Surgery (1); Radiofrequency Ablation (1); Soft Tissue Ablation (1); Trigger Finger Surgery (1)
Tremor (Nervous system disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Viremia (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT03533946/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT03533946/ICF_002.pdf